CLINICAL TRIAL: NCT06154733
Title: MANAGEMENT OF HYPERSENSITIVITY IN MOLAR INCISOR HYPOMINERALISATION USING LOW LEVEL LASER IN CHILDREN (RANDOMIZED CLINICAL TRIAL)
Brief Title: HYPERSENSITIVITY IN MOLAR INCISOR HYPOMINERALISATION USING LOW LEVEL LASER IN CHILDREN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Baraka, Lecturer, Pediatric dentistry department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0774-09/2023
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-09

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralisation, Low Level Laser, Sealant, Hypersensitivity
MeSH Terms: conditions — Molar Hypomineralization; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: All selected first permanent molars will be randomly equally allocated into three groups. Group 1(n=15): PBM with LLLT, Group 2 (n=15): Resin-based sealant (Fissured Nova Plus) and Group 3 (n=15): Glass ionomer sealant (Ketac).
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of examiners is impossible to be done during intervention due to different natures of the materials. However, the evaluator at follow-up visits, patients and the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Photobiomodulation with low level laser therapy (Experimental): This group will be subjected to photo biomodulation by low level laser therapy. Diode laser will be used (SIROLaser Blue®, Sirona, Germany) at a wavelength of 660 nm and a power of 100 mW for 10 sec, corresponding to an energy dose of 1 J. Irradiation will be performed at the hypomineralized area: two irradiations scanning the surface in the mesiodistal direction and two in the occlusogingival direction (perpendicular to the tooth surface) precisely over the lesion, in a uniform scanning motion with relative isolation. Treatment will be performed in 3 sessions with a 72-hour interval between sessions. During the laser treatments, both the volunteer and operator will use protective eyewear and all rules of safety will be obeyed.
  Interventions: Procedure: Photobiomodulation usinf low level laser therapy
- light cured resin-based sealant (Active Comparator): This group will receive light cured resin-based sealant (Fissured Novo Plus). Cotton rolls and a four-handed technique will be applied for isolation. Scotchbond Universal will be rubbed in the cleaned surface for 20 seconds and air dried for 5 seconds. Afterwards, Fissured Novo Plus will be applied with a syringe. Before light-curing, the presence of air bubbles will be checked and teased out. Light curing for 40 seconds will be done. Occlusion will be checked using articulating paper and necessary adjustments will be done using finishing burs.
  Interventions: Procedure: Resin-based sealant
- glass ionomer sealant (Active Comparator): This group will receive glass ionomer sealant. Fuji triage will be applied after activating and mixing the capsule. Light cure for 20 seconds. Occlusion will be checked using articulating paper and necessary adjustments will be done using finishing burs.
  Interventions: Procedure: Glass ionomer sealant

INTERVENTIONS:
Procedure: Photobiomodulation usinf low level laser therapy — Diode laser will be used (SIROLaser Blue®, Sirona, Germany) at a wavelength of 660 nm and a power of 100 mW for 10 sec, corresponding to an energy dose of 1 J. Irradiation will be performed at the hypomineralized area: two irradiations scanning the surface in the mesiodistal direction and two in the occlusogingival direction (perpendicular to the tooth surface) precisely over the lesion, in a uniform scanning motion with relative isolation. Treatment will be performed in 3 sessions with a 72-hour interval between sessions.
  Arms: Photobiomodulation with low level laser therapy
Procedure: Resin-based sealant — Cotton rolls and a four-handed technique will be applied for isolation. Scotchbond Universal will be rubbed in the cleaned surface for 20 seconds and air dried for 5 seconds. Afterwards, Fissured Novo Plus will be applied with a syringe. Before light-curing, the presence of air bubbles will be checked and teased out. Light curing for 40 seconds will be done. Occlusion will be checked using articulating paper and necessary adjustments will be done using finishing burs.
  Arms: light cured resin-based sealant
Procedure: Glass ionomer sealant — Fuji triage will be applied after activating and mixing the capsule. Light cure for 20 seconds. Occlusion will be checked using articulating paper and necessary adjustments will be done using finishing burs.
  For the duration of the study, children will be instructed to undergo regular tooth brushing and flossing. Any other needed treatment will be done for the child.
  Arms: glass ionomer sealant

SUMMARY:
Molar Incisor Hypomineralisation (MIH) is a qualitative defect of enamel that shows asymmetrically involvement of one to four on first permanent molars (FPM) with or without incisor teeth involvement. Hypersensitivity is one of the biggest challenges in the treatment of MIH. A sample of children having a first permanent molar erupted with MIH and suffering of dentin hypersensitivity (DH). All selected 45 first permanent molars will be randomly equally allocated into three groups. DH will be evaluated after the treatments. The primary outcome of this study is change in pain/sensitivity, when evaluated through a Visual Analogue Scale. OHRQoL will be also assessed for all children through the child perceptions questionnaire (CPQ8-10).

DETAILED DESCRIPTION:
Background: Molar Incisor Hypomineralisation (MIH) is a qualitative defect of enamel that shows asymmetrically involvement of one to four on first permanent molars (FPM) with or without incisor teeth involvement. Hypersensitivity is one of the biggest challenges in the treatment of MIH.

Aim of the study: To evaluate the effectiveness of photo biomodulation (PBM) with low-level laser therapy (LLLT) in the management of hypersensitivity in children diagnosed with MIH in comparison to resin-based fissure sealant (Fissured Novo Plus) and glass ionomer sealant (Ketac) and the impact of LLLT on their oral health-related quality of life (OHRQoL).

Materials and Method: A sample of children with an age range of 8-10 years old, having a first permanent molar erupted with MIH and suffering of dentin hypersensitivity (DH), will be selected from the outpatient clinic of Pediatric Dentistry and Public Health Department, Faculty of Dentistry, Alexandria University after securing necessary consents. All selected 45 first permanent molars will be randomly equally allocated into three groups. Group 1(n=15): PBM with LLLT, Group 2 (n=15): Resin-based sealant (Fissured Nova Plus) and Group 3 (n=15): Glass ionomer sealant (Ketac). DH will be evaluated 15 min after the application of the treatments and the patients will be reevaluated 1 week, 1 month, 3 months and 6 months after the treatments. The primary outcome of this study is change in pain/sensitivity, when evaluated through a Visual Analogue Scale, to determine the effectiveness of the proposed treatments, as well as differences among the evaluation times for each proposed treatment. OHRQoL will be also assessed for all children through the child perceptions questionnaire (CPQ8-10) which will be administered at the beginning and the end of the treatment.

Results: The data will be collected, tabulated, and analyzed using suitable statistical tests to achieve the aim of the study.

ELIGIBILITY:
Inclusion Criteria:

* 6-10-year-old children (15).
* At least one tooth with MIH and DH reported in the occlusal region with sensitivity equal to or greater than 4 on the Visual analogue Scale (VAS).
* Good overall health (ASA I).

Exclusion Criteria:

* First permanent molars with active carious lesions or defective restorations
* Sufficient dentin loss that requires restorative therapy.
* Any clinical signs of failure (abscess, fistula).
* Patients with systemic diseases.
* Having undergone any professional desensitizing treatment in the previous 6 months.
* Having used a desensitizing paste in the previous 3 months.
* Use of anti-inflammatory drugs or analgesics at the time of recruitment.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Dentin Hypersensitivity | Day0, 1 week, 1 month, 3 months and 6 months
  it will be measures usinf a Faces pain scale

SECONDARY OUTCOMES:
Oral health related Quality of life (OHRQoL) | Day 0
  OHRQoL will be assessed for all children through the validated Arabic version of the Child Perceptions Questionnaire (CPQ8-10)which will be administered at the beginning and the end of the treatment. The questionnaire evaluates the severity of oral symptoms, functional limitations as well as emotional and social well-being. The questions are measured using a 5-point Likert scale as follows: never = 0, once or twice = 1, sometimes = 2, often = 3, and Every day or almost every day = 4. Hence, total scores range from 0 to100, and higher scores indicate poorer OHRQoL.

IPD SHARING:
Plan to Share IPD: Undecided